CLINICAL TRIAL: NCT01663389
Title: An Open Label, Non-Randomized, Single Dose, Two Period, Cross-Over, Mass Balance Study to Investigate the Recovery, Excretion, and Pharmacokinetics of 14C -GSK1322322 Administered as a Single Intravenous and Single Oral Dose to Healthy Adult Male Subjects
Brief Title: A Study to Investigate the Recovery, Excretion, and Pharmacokinetics of 14C -GSK1322322 After an Intravenous and an Oral Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 112167
Record Dates: First submitted 2012-07-19; First posted 2012-08-13 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Infections, Bacterial
Keywords: mass balance; radiolabel; oral; IV; GSK1322322; healthy volunteer; antibiotic
MeSH Terms: conditions — Bacterial Infections | interventions — GSK1322322

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1322322 1000 mg IV (Experimental): On Day 1 of Period 1, after an overnight fast, subjects will receive GSK1322322 1000 mg IV single dose (containing approximately 45.5 microcurie [μCi] radioactive 14C-GSK1322322) for intravenous infusion over 60 minutes.
  Interventions: Drug: GSK1322322 1000 mg containing radioactive 14C-GSK1322322
- GSK1322322 1200 mg Oral Solution (Experimental): On Day 1 of Period 2, after an overnight fast, subjects will receive GSK1322322 1200 mg oral solution single dose (containing approximately 54.5 μCi radioactive 14C-GSK1322322).
  Interventions: Drug: GSK1322322 1200 mg containing radioactive 14C-GSK1322322

INTERVENTIONS:
Drug: GSK1322322 1000 mg containing radioactive 14C-GSK1322322 — GSK1322322 1000 mg is a mesylate salt powder for injection containing 45.5 μCi radioactive 14C-GSK1322322 1000 mg as free base.
  Arms: GSK1322322 1000 mg IV
Drug: GSK1322322 1200 mg containing radioactive 14C-GSK1322322 — GSK1322322 1200 mg is a mesylate salt powder for oral solution containing 54.5 μCi radioactive 14C-GSK1322322 1200 mg as free base.
  Arms: GSK1322322 1200 mg Oral Solution

SUMMARY:
This is a phase 1, non-randomized, open label, single-dose, two-period, cross-over study. This study will utilize 14C radiolabeled GSK1322322 to investigate the recovery, excretion, and pharmacokinetics of GSK1322322 in 6 healthy adult male subjects through the sampling of blood, urine, and feces.

Each subject will participate in the study for approximately 7 to 8 weeks i.e., 30 day screening period, two dosing periods (approximately 8 days each) and a follow up visit.

The subjects will be admitted to the clinical unit on Day 1 of the first treatment period and remain in the unit for up to approximately 16 days through the end of the second treatment period.

On Day 1 of Period 1, each subject will receive 14C radiolabeled GSK1322322 as a single therapeutic intravenous (IV) dose (1000 milligrams [mg]). When the total radioactivity is <1% of the administered dose in all subjects, Period 2 dosing will begin (approximately 8 days after the IV dose). On Day 1 of Period 2, each subject will receive single therapeutic oral solution dose (1200 mg). Blood, urine, bile and fecal samples will be collected during both the periods. The subject may be discharged from the unit as early as Day 8 of Period 2. Subjects will visit the study unit for the follow-up visit 7 to 10 days following discharge from the unit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 30 and 55 years of age, with body weight between 60 to 80 kilograms (kg) and a history of regular bowel movements
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods from first dose of study medication until the final follow up visit
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin =<1.5x upper limit of normal
* QT interval by Bazett's correction formula (QTcB) <450 millisecond (msec); or QTcB <480 msec in subjects with Bundle Branch Block
* Available to complete the study and return for follow-up visits if necessary
* Capable of giving written informed consent

Exclusion Criteria:

* Any condition that could interfere with the accurate assessment and recovery of radioactivity [14C]
* Participation in a clinical trial involving administration of radiolabeled 14C-labelled compound(s) within the last 12 months
* Any condition which impairs the absorption, distribution, metabolism or excretion of the investigational product
* Subjects with a history of cholecystectomy
* Subject has received a total body radiation dose of greater than 5.0 millisievert (mSv) or exposure to significant radiation during 1 year before dosing
* The subject has a positive: drug/alcohol, Hepatitis, HIV screen
* Abuse of alcohol
* History of liver disease, or known hepatic or biliary abnormalities
* The subject has recently received an investigational product
* Donation of more than 500 mL blood within a 56 day period
* Unwillingness or inability to follow the procedures outlined in the protocol
* Use of prescription or non-prescription drugs
* Subject is mentally or legally incapacitated
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Smoking or history or regular use of tobacco or nicotine-containing products
* Unable to refrain from consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose
* History of cardiac disease

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-08-10 (Actual); Primary Completion 2012-10-05 (Actual); Study Completion 2012-10-05 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters of GSK1322322 and radiolabeled compound following single IV or oral solution dose: AUC(0-infinity), AUC(0-t), Cmax, tmax, t1/2 for IV and oral solution regimens and CL and Vss for IV regimen only | Day 1 through Day 8 of Period 1 and Period 2 (16 days)
  Plasma PK parameters will be statistically summarized by treatment. Plasma concentration-time data will be analyzed by non-compartmental methods. Following PK parameters will be studied: Area under the concentration-time curve (AUC) from time zero (pre-dose) extrapolated to infinite time [AUC(0-infinity)], AUC(0-t), maximum observed concentration (Cmax), time of occurrence of Cmax (tmax), terminal phase half-life (t1/2) for IV and oral solution regimens and systemic clearance (CL) and volume of distribution (Vss) for IV regimen only.
Percent total recovery of radioactivity in urine and feces in each interval and cumulative | Day 1 through Day 8 (and additional days, if required) of Period 1 and Period 2 (16 days or more)
  Total recovery of radioactivity in urine and feces (as a percentage of total radioactive dose in each interval and cumulative)

SECONDARY OUTCOMES:
Safety parameters including adverse events, clinical laboratory tests, concomitant medications, electrocardiograms, and vital signs | Duration of the study (56 days)
  To evaluate the safety and tolerability of GSK1322322 after single IV and oral solution doses in healthy subjects safety parameters will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 112167 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112167?search=study&search_terms=112167#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 112167 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112167 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112167 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112167 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112167 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112167 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112167 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register